CLINICAL TRIAL: NCT04188093
Title: Identifying Patients in Risk of Post-operative Complications Using PACU Discharge Criteria and Need for Interventions in the PACU Setting
Brief Title: Identifying Patients in Risk of Post-operative Complications Using PACU Discharge Criteria
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Eske Kvanner Aasvang, Head of research, Clinical professor, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: PIRCPAC
Record Dates: First submitted 2019-11-26; First posted 2019-12-05 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Complication,Postoperative; Post-Op Complication
Keywords: PACU; Postoperative Care Unit; Continous monitoring; PACU discharge criteria
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PACU discharge criteria and continuous monitoring on the ward — * PACU discharge criteria (modified aldrete score).
  * Continous monitoring of vital signs 96 postoperative hours

SUMMARY:
In the Postoperative Care Unit surgical patients are monitored closely to ensure safe condition before transfer to the ward. This study will aim to identify patients in risk of complications on the ward using the national postanesthesia care unit (PACU) discharge criteria, a modified Aldretes score. Secondary to identify patients in risk of micro events as detected by continuous monitoring of vital signs on the ward.

DETAILED DESCRIPTION:
Patients undergoing esophageal resection and pancreaticoduodenectomy are at high risk of developing complications after surgery. Described patient groups are monitored for at least 24 hours in PACU before returning to the ward.

In Denmark physiological parameters are assessed in the PACU every hour until discharge using the DASAIM discharge criteria (A modified Aldrete score).

The PACU discharge score is calculated on parameters including sedation, respiratory rate, saturation, systolic blood pressure, puls, physical capability (if epidural or spinal anesthesia), pain in rest, nausea, diuresis and temperature. Each parameter is given a score between 0 and 3. 0 describes no problem and 3 describes a severe problem.

The investigators will investigate the predictive value of the PACU discharge criteria and interventions in the PACU setting, to identify patients at risk of developing postoperative complications. Secondary outcome is micro events on the ward. Patients vital signs are monitored continuously from PACU discharge until the 5th postoperative day. Micro events are defined as deviations of vital parameters from normal range.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* Pancreaticoduodenectomy (KJLC30)
* Transthoracic esophageal resection without interposition (KJCC10)

Exclusion Criteria:

* Patients not expected to be able to cooperate
* Patients not cognitive well (Mini Mental State Examination < 24)
* Pacemaker
* Patients with allergies including band aid, plastic and silicone

Ages: 60 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients over 60 years under surgery for abdominal cancer.
  * Pancreaticoduodenectomy (KJLC30)
  * transthoracic esophageal resection without interposition (KJCC10)
  Patients undergoing described surgery stay at least 24 hours in PACU following local guidelines
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Clinical in-hospital complications | until discharge, up to 90 days
  Occurence of clinical complications occuring during the hospital stay (pneumonia, myocardial infarction, brain stroke, renal impairment, etc), based upon international definitions

SECONDARY OUTCOMES:
Bradycardia | During the first 4 postoperative days
  pulse <40/min measured by pulse oximeter
Tachycardia | During the first 4 postoperative days
  pulse >140/min meausured by pulseoximetry
Severe desaturation | During the first 4 postoperative days
  Arterial saturation <85% lasting >10 minutes per episode, measured by pulse oximeter
Very severe desaturation | During the first 4 postoperative days
  Arterial saturation <80% lasting >10 minutes per episode, measured by pulse oximeter
Hypotension | During the first 4 postoperative days
  Middle arterial blood pressure <75 for >29 minutes measured by non-invasive manometer
Severe hypotension | During the first 4 postoperative days
  Middle arterial blood pressure <65 for >29 minutes measured by non-invasive manometer
bradypnea | During the first 4 postoperative days
  respiratory rate <8/min for 30 minutes, measured by ECG
Tachypnea | During the first 4 postoperative days
  respiratory rate >20/min for 30 minutes, measured by ECG
Severe tachypnea | During the first 4 postoperative days
  respiratory rate >30/min for 30 minutes, measured by ECG
Clinical out of hospital complications | until 96 days postoperatively
  Occurence of clinical complications occuring after the hospital stay (pneumonia, myocardial infarction, brain stroke, renal impairment, etc), based upon international definitions

OTHER OUTCOMES:
description of other physiological deviations | during hospital stay, up to 30 days
  description og frequency and duration of other physiological deviations (fever, arrythmia, apnea, arrythmia, etc)

CONTACTS AND LOCATIONS:
Overall Officials: Eske K Aasvang, Dr. Med., Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided